CLINICAL TRIAL: NCT00180037
Title: Multicenter, Placebo Controlled, Randomized, Double-Blinded Study: Coenzyme Q10 Nanodispersion Versus Placebo as Symptomatic Treatment in Parkinson's Disease
Brief Title: Coenzyme Q10 as a Symptomatic Treatment in Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Deutsche Parkinson-Vereinigung e.V. (Unknown); MSE Pharmazeutika GmbH, Bad Homburg (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 78052003
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2009-01-19 (Estimated); Status verified 2009-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Coenzyme Q10; Treatment; Neuroprotection
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Coenzyme Q10 Nanodispersion (Nanoquinone)
Drug: Placebo

SUMMARY:
This study was designed to evaluate the symptomatic effects of Coenzyme Q10 nanodispersed solution in middle-stage Parkinson's disease (PD) patients (Hoehn&Yahr II to III). The treatment phase includes three months period of 300 mg Coenzyme Q10 per day or placebo.

The primary outcome measure was the combined Unified Parkinson's Disease Rating Scale (UPDRS) Part II and III.

The hypothesis of this study was that Coenzyme Q10 improves the energy status of the diseased dopaminergic neuronal cell type and thus producing more dopamine leading to an improvement of parkinsonian symptoms in PD patients.

DETAILED DESCRIPTION:
This study was designed to evaluate the symptomatic effects of Coenzyme Q10 nanodispersed solution in middle-stage non-fluctuating Parkinson's disease (PD) patients (Hoehn&Yahr II to III). The treatment phase includes three months period of 300 mg Coenzyme Q10 per day or placebo.

The design of the study was a prospective, randomized, multicenter, double-blind placebo-controlled protocol. The intervention includes 100 mg Coenzyme Q10 nanodispersion (Nanoquinon solution) tid or matched placebo for three months.

Participating study centers include Neurological University Outpatient Clinics and Neurological Departments of Community-based Hospitals experienced with PD patients.

The primary outcome measure was the combined Unified Parkinson's Disease Rating Scale (UPDRS) Part II and III.

The hypothesis of this study was that Coenzyme Q10 improves the energy status of the diseased dopaminergic neuronal cell type and thus producing more dopamine leading to an improvement of parkinsonian symptoms in PD patients.

Main inclusion criteria:

* Parkinson's disease according to the UK Brain Bank criteria
* Hoehn & Yahr stadium II until III
* Age 40 to 75 years
* UPDRS Part III > 15 points
* No motor fluctuations or dyskinesias
* Stable medication for 4 weeks prior to inclusion

Main exclusion criteria:

* Atypical parkinsonian syndromes
* Dyskinesias or motor fluctuations
* Coenzyme Q10 treatment in the past
* Pregnancy

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease according to the UK Brain Bank criteria
* Hoehn & Yahr stadium II until III
* Male or female
* Age 40 to 75 years
* UPDRS Part III > 15 points
* No motor fluctuations or dyskinesias
* Stable parkinsonian condition for 4 weeks prior to inclusion
* Outpatients
* Patients without or with stable levodopa treatment for 4 weeks prior inclusion
* Written informed consent

Exclusion Criteria:

* Atypical or drug-induced parkinsonian syndromes
* Dyskinesias or motor fluctuations
* Coenzyme Q10 treatment in the past
* Pregnancy
* Epileptic seizures in the history
* Hypothyroidism
* Severe medical conditions with interference with study drug
* Treatment with CSE inhibitors, thyroidal hormones, antiarrhythmic drugs, warfarin, metformin
* Treatment or intake of vitamins, magnesium, vitamin E, calcium

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132
Dates: Start 2003-09; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) Part II and III

SECONDARY OUTCOMES:
Total UPDRS
Safety
PDQ-39
SF36
CGI
Schwab&England
Montgomery-Asperg
Pain
Incontinence
Sexual behavior

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Reichmann, MD, Principal Investigator — Technical University of Dresden
Locations (13):
- Germany (13):
  - Department of Neurology, University of Ulm, Ulm, Baden-Wurttemberg
  - Department of Neurology, Fachklinik Ichenhausen, Ichenhausen, Bavaria
  - Department of Neurology, Leopoldina Krankenhaus, Schweinfurt, Bavaria
  - Department of Neurology, University of Marburg, Marburg, Hesse
  - Department of Neurology, Deutsche Klinik fuer Diagnostik, Wiesbaden, Hesse
  - Department of Nuerology, Klinikum Lippe, Lemgo, Lower Saxony
  - Department of Neurology, Klinikum Lueneburg, Lüneburg, Lower Saxony
  - Department of Neurology, Ruhr-University of Bochum, Bochum, North Rhine-Westphalia
  - Department of Neurology, Klinikum Essen-Borbeck, Essen, North Rhine-Westphalia
  - Department of Neurology, Klinik Ambrock, Hagen, North Rhine-Westphalia
  - Department of Neurology, University of Homburg, Homburg, Saarland
  - Department of Neurology, Technical University of Dresden, Dresden, Saxony
  - Department of Neurology, Charite Berlin, Berlin, State of Berlin

REFERENCES:
- [Result] Storch A, Jost WH, Vieregge P, Spiegel J, Greulich W, Durner J, Muller T, Kupsch A, Henningsen H, Oertel WH, Fuchs G, Kuhn W, Niklowitz P, Koch R, Herting B, Reichmann H; German Coenzyme Q(10) Study Group. Randomized, double-blind, placebo-controlled trial on symptomatic effects of coenzyme Q(10) in Parkinson disease. Arch Neurol. 2007 Jul;64(7):938-44. doi: 10.1001/archneur.64.7.nct60005. Epub 2007 May 14. PMID 17502459
- See also: Homepage of Principle study center — http://www.neuro.med.tu-dresden.de